CLINICAL TRIAL: NCT04468724
Title: MAKASI. An Intervention for African and Caribbean Migrants' Empowerment in Sexual Health in Order to Reduce Their Social and Health Vulnerabilities in Paris Greater Area
Brief Title: MAKASI Intervention for African and Caribbean Migrants' Empowerment in Sexual Health in Paris Greater Area
Acronym: MAKASI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Agence Regionale de Sante d'Ile de France (Other Government)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 14056
Record Dates: First submitted 2020-06-26; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: HIV/AIDS; STI
Keywords: Migrants; Sexual Health; Empowerment; community-based intervention; HIV prevention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Empowerment

STUDY DESIGN:
Intervention Model Description: In order to measure the impact of the intervention, we propose a two-arm essay: an intervention arm and a control arm. However, for ethical reasons, it was impossible not to offer help to all the screened persons who were in need of help for social or health reasons. That is why we will compare an arm where the intervention is immediate with an arm where the intervention is differed by three months (control arm). The comparison about what happens in the three first months will allow us to measure the impact of the intervention at three months. All participants will have a follow up of six months after the intervention.
  The participants will be randomly allocated to the immediate arm or the differed arm (please see below).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMMEDIATE (Experimental): People who are included in the Immediate Arm receive the Makasi intervention right away or in a six-week time if they are not available on the spot
  Interventions: Behavioral: MAKASI
- DIFFERED (Other): People who are included in the Differed Arm receive the Makasi intervention three months after inclusion
  Interventions: Behavioral: MAKASI

INTERVENTIONS:
Behavioral: MAKASI — The Makasi intervention consists in a unique Empowerment interview, based on motivational interviewing techniques. Is is made of three components:
  * Listening and building trust
  * Active referral to structures that answers sanitary and social needs
  * Sexual Health Prevention
  Materials used are: referral letters, bilingual health guides, adapted maps of the the neighborhoods with useful addresses.
  The Makasi intervention is proposed and delivered in an outreach setting: health mediators propose information on general health and rapid HIV and HCV testing. They screen the people attending and propose Makasi to eligible persons.

SUMMARY:
Background. Immigrants from Sub-Saharan Africa are the second group most affected by HIV in France. Part of these HIV infections occurred after arrival in France, in relation to social hardships. Immigrants coming from the non-French Caribbean islands face similar difficulties. Many actors strive for an easier access to healthcare services for immigrants; however the mere supply of knowledge and medicalised solutions is not enough to make persons adopt prevention behaviours. It seems necessary to act upon empowerment to bring resources to individuals and communities in order to improve their autonomy and action capacity. Civil Society Organisations and researchers join forces in the MAKASI interventional research which aims at reinforcing immigrants' empowerment in sexual health in order to reduce their exposure to sexual risks.

Objectives : The MAKASI intervention consists in a unique Empowerment interview based on the principles of motivational interviewing, using an Active Referral system to social or sanitary services relevant to the person's needs. Our hypothesis is that this intervention is going to reinforce four dimensions of empowerment in sexual health among immigrants: the capacity to express their needs, competencies in sexual, self-esteem, awareness of exposure to HIV and STIs. The proposed research aims at measuring the efficacy of the intervention on these four dimensions, and at evaluating its processes and efficiency (cost-efficacy).

Methods: The intervention is delivered within the mobile units of Afrique Avenir in the public spaces where African and Caribbean populations live and work. The evaluation uses integrated mixed-method approach, combining a quantitative evaluation of impact and a qualitative research on processes. The measure of impact will be done by comparing indicators on the four dimensions of empowerment in sexual health and indicators of exposure to sexual risks, between an arm where the intervention is immediate and an arm where the intervention is differed by 3 months (control arm). The qualitative evaluation of the intervention processes will be based upon an ethnographic approach of the intervention and the participants' experience.

Perspectives: This project will demonstrate the efficacy and the efficiency of an innovative intervention aiming at reducing Sub-Saharan and Caribbean immigrants' exposure to risks in sexual health.

DETAILED DESCRIPTION:
Migrants from Sub-Saharan Africa are the second group most affected by HIV epidemic in France. Previous study established that part of HIV infections among Sub-Saharan migrants occurred after arrival in France, and that the exposure to sexual risks was linked both to social hardships and structural difficulties experienced during the settlement period in France. Many actors strive for an easier access to healthcare services for migrants, however the mere supply of knowledge and medicalised solutions is not enough to make persons adopt protection or healthcare practices. It seems necessary to work for the individual and community empowerment in order to bring resources to individuals and communities so they can more easily take action in the new and complex context of a host country.

To improve the prevention of sexual risks in this population coming from Sub-Saharan Africa, local charities and researchers join forces in order to propose an interventional research which aims at enabling Sub-Saharan migrants to appropriate prevention and healthcare means, especially in the area of sexual health, to reinforce their autonomy, their capacity and power to take action and to protect their health against the disruption caused by migration and the difficulty in accessing rights and fundamental needs.

The pilot phase of this research has made it possible to build an empowerment intervention which consists of a single individual interview based on the principles of motivational maintenance, articulated with an active orientation towards adequate social or health services, possibly accompanied when necessary. Our hypothesis is that this intervention will strengthen four dimensions of empowerment in sexual health among immigrants:

* Ability to express needs: Ability to talk about sexuality or sexual health to peers or professionals
* sexual health skills: know the different tools of combined prevention, know where to go for screening, gynaecology or sexual health consultation
* self-esteem: knowing your rights, having the material means (housing, administrative situation, financial resources) to refuse a situation of sexual constraint and avoid being exposed to violence, feeling that you can act on your own situation (sense of personal effectiveness)
* awareness of HIV exposure and its determinants: being informed about the epidemiology of HIV, the fact that it is possible to be infected in France, and risk factors

Objectives

To strengthen the sexual health empowerment of immigrants from sub-Saharan Africa and the Caribbean, we propose to act on the four dimensions of sexual empowerment with the following specific objectives:

Ability to express needs:

* Speaking up
* Reduce social isolation

Sexual Health Skills:

* Improve knowledge of health and social resources
* Improve access to screening
* Improve access to sexual health services (Contraception, condoms, Prep)
* Improve ownership of combined prevention

Self-esteem:

* Improve people's autonomy in social processes (housing, paper)
* Improving Mental Health: Reducing Psychological Distress and Suffering
* Improve personal efficiency

Awareness of HIV and STI exposure

• Improve perception of HIV and STI exposure, effectiveness of antiretroviral treatment and preventive strategies.

The research aims to measure the effectiveness of the intervention against all of these indicators, as well as to conduct an evaluation of the processes and efficiency (cost-effectiveness).

Methods:

The intervention is part of the action already carried out by the mobile team of Afrique Avenir, which offers in strategic places of passage (markets, squares, RER stations, etc.) an awareness of sexual health through cultural mediation and a TROD offer. The MAKASI intervention involves identifying immigrants in precarious situations and exposed to HIV in these awareness-raising places, offering them a personalized interview with a health mediator to help them prioritize their needs, and guide them through the health and welfare system.

To assess this complex intervention, we will use an integrated mixed-method approach. A quantitative impact assessment and a qualitative assessment of the processes will be conducted in parallel to establish, by integrating these data, the causal attribution of the effects of the intervention.

Quantitative assessment of impact:

To measure the impact of the intervention, we propose a two-arm diagram: an intervention arm and a control arm. However, for ethical reasons, in order to offer help to all identified people with social or health needs, we will compare an arm where the intervention is immediate, and an arm where it is delayed by 3 months (control arm). The comparison of what happens in the first three months will measure the short-term effect of the intervention, and establish a causal link between the intervention and the observed changes. All people, in both arms, will be followed six months to observe the evolution of the indicators in the medium term. The impact assessment of the intervention will be made possible both by comparison between the immediate intervention arm and the control arms in the first three months, and by comparison before/after the intervention in both arms). Individuals will be randomly allocated to the immediate or delayed intervention arm after an initial interview to identify social and health needs. The goal is to include 1200 people (600 in each arm).

Qualitative assessment of processes and effects:

The qualitative analysis of the processes aims to highlight and analyse the successes, failures and limitations of the intervention, with particular regard to the implementation and its effects. It will also be necessary to produce knowledge on the conditions of reproduction or the extension of the intervention. This analysis will be based on an ethnographic approach to the intervention and the participants' journey, with a work of observation of the different stages and in-depth and repeated semi-directive interviews.

Cost collection will measure the efficiency of the response.

Expected results :

This project will demonstrate the effectiveness and efficiency of an innovative intervention to reduce exposure to sexual health risks among immigrants from sub-Saharan Africa and the Caribbean, and will highlight the conditions of its reproduction or extension. It is closely linked to the initiative towards Paris without AIDS, which develops the collective dimensions of empowerment through different approaches in the communities concerned.

ELIGIBILITY:
Inclusion Criteria:

* Be aged at least 18
* HIV negative
* Born in sub-Saharan Africa or the non-French Carribean
* At least one of the eight vulnerability criteria: no stable house, no job, food deprivation, no papers, feeling isolated, not knowing where to go to to the doctor, no health insurance, experiencing violence

Exclusion Criteria:

* Does not speak French or English
* Persons whose rapid HIV or HCV test is reactive
* Persons who are not able to give an informed consent: bad mental health, persons who are on drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Change of unprotected sex | 0, 3 months, 6 months after inclusion
  Declare unprotected sex at least once during the last three months (percent)
Change of transactional sex | 0, 3 months, 6 months after inclusion
  Declare Transactional sex at least once during the last three months (percent)
Change of Forced sex | 0, 3 months, 6 months after inclusion
  Declare having forced to have sex at least once during the last three months (percent)

SECONDARY OUTCOMES:
Empowerment - Social Isolation | 0, 3 months, 6 months after inclusion
  Feeling to be alone (percent)
Empowerment - Ability to talk | 0, 3 months, 6 months after inclusion
  Empowerment - Perception of ability to talk about one's situation with a professional (percent)
Empowerment - Health insurance | 0, 3 months, 6 months after inclusion
  Empowerment - having a health insurance (percent)
Empowerment - HIV test | 0, 3 months, 6 months after inclusion
  Empowerment - Has been HIV tested
Empowerment - TASP knowledge | 0, 3 months, 6 months after inclusion
  Empowerment - Knowledge that HIV treatment prevents from transmitting HIV
Empowerment - mental health score | 0, 3 months, 6 months after inclusion
  Empowerment - PHQ 9 (Patient Health Questionnaire in 9 items) score : from 0 (good mental health) to 9 (very bad mental health)
Empowerment - self-efficacy | 0, 3 months, 6 months after inclusion
  Empowerment - feeling of control over the decisions that affect its life (percent)
Empowerment - HIV risk awareness | 0, 3 months, 6 months after inclusion
  Empowerment - knowing that the risk of being HIV infected concerns everyone (percent)
Empowerment - access to healthcare structure | 0, 3 months, 6 months after inclusion
  Empowerment - having had access to a health structure when needed, in the last 3 months (percent)

CONTACTS AND LOCATIONS:
Overall Officials: Annabel Desgrées du Loû, PhD, Principal Investigator — French Institute for Sustainable Developement (IRD)
Locations (1):
- Afrique Avenir Mobile Unit, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gosselin A, Carillon S, Coulibaly K, Ridde V, Taeron C, Kohou V, Zoumenou I, Mbiribindi R, Derche N, Desgrees du Lou A; MAKASI Study Group. Participatory development and pilot testing of the Makasi intervention: a community-based outreach intervention to improve sub-Saharan and Caribbean immigrants' empowerment in sexual health. BMC Public Health. 2019 Dec 5;19(1):1646. doi: 10.1186/s12889-019-7943-2. PMID 31805909
- [Derived] Coulibaly K, Gosselin A, Derche N, Mbiribindi R, Desgrees du Lou A; MAKASI Study Group. Association between HIV risk perception, knowledge of biomedical prevention and sexual behaviour among sub-Saharan African immigrants living in a precarious situation in France. Sex Transm Infect. 2025 Jul 17;101(5):294-300. doi: 10.1136/sextrans-2024-056392. PMID 39884844
- [Derived] Goncalves Tasca B, Bousmah MA, Coulibaly K, Gosselin A, Ravalihasy A, Desgrees du Lou A, Melchior M; Makasi Study Group. Depression and loneliness among Sub-Saharan immigrants living in the greater Paris area: results from the MAKASI empowerment stepped wedge cluster randomised controlled trial. Soc Psychiatry Psychiatr Epidemiol. 2024 Nov;59(11):2049-2061. doi: 10.1007/s00127-024-02665-7. Epub 2024 Apr 7. PMID 38584200
- [Derived] Coulibaly K, Bousmah MA, Ravalihasy A, Taeron C, Mbiribindi R, Senne JN, Gubert F, Gosselin A, Desgrees du Lou A; MAKASI Study Group. Bridging the knowledge gap of biomedical HIV prevention tools among sub-saharan african immigrants in France. Results from an empowerment-based intervention. SSM Popul Health. 2023 Jul 23;23:101468. doi: 10.1016/j.ssmph.2023.101468. eCollection 2023 Sep. PMID 37560089